CLINICAL TRIAL: NCT03619707
Title: Oral Dydrogesterone Versus Vaginal Progesterone in the Luteal Phase Support in Cryo-warmed Embryo Transfer Cycles: Randomized Controlled Trial
Brief Title: Oral Versus Vaginal Progesterone in the Luteal Support in Cryo-warmed Embryo Transfer Cycles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Johnny Awwad, Professor of Obstetrics and Gynecology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AmericanUBMC-CWET
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Sterility; Infertility
Keywords: Luteal Phase Support; Cryo-warmed Embryo Transfer; Assisted Reproductive Technology
MeSH Terms: conditions — Infertility | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Dydrogesterone (Experimental): Oral dydrogesterone (Duphaston 10 mg) will be given orally four times daily : will be continued till the pregnancy test, and till at least 12 weeks of gestation in case of a positive pregnancy test.
  Interventions: Drug: Progesterone
- Vaginal microprogesterone (Experimental): Vaginal progesterone (Utrogestan 200 mg) will be given vaginally four times daily: will be continued till the pregnancy test, and till at least 12 weeks of gestation in case of a positive pregnancy test
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — Patients will be randomly assigned during the treatment follow up, at the time of addition of progesterone to the regimen, following computerized random number generator in procedure, to one of the study groups. Patients will be aware of the allocated arm since the treatment drugs have different route of administration. Group I will receive the oral dydrogesterone, while group II will receive the vaginal microprogesterone.

SUMMARY:
In IVF/ICSI cycles, the progesterone levels induced by ovarian stimulation are low, therefore the luteal phase is supported by progesterone. The use of progestogens in IVF is associated with an improvement in the live birth rate Standard protocol for luteal phase support has not yet been established. Currently vaginal progesterone is widely used, since the classic oral progesterone seems to result in a low bioavailability and a lower pregnancy rate. However, vaginal administration of progesterone is associated with vaginal irritation, discharge and bleeding. For all these reasons, there is a need for an effective, well tolerated, and safe treatment that can improve patient satisfaction and compliance.

Many studies have observed similar pregnancy rate results with dydrogesterone and micronized vaginal progesterone. A new RCT including a total of 1143 patients by Tournaye, showed that dydrogesterone treatment had a similar safety profile to micronized vaginal progesterone (MVP) for luteal support as part of ART treatment. The crude pregnancy rates at 12 weeks were 37.6% and 33.1% in the dydrogesterone and MVP treatment groups respectively.

Regarding the administration route of progesterone, intramuscular and transvaginal routes are the two conventional progesterone administration techniques. However, very few studies have compared the advantages of oral dydrogestrone with vaginal progesterone for luteal support in ART cycles.

The objective of the investigator's study is to demonstrate the superiority of oral dydrogesterone (Duphaston) 10 over MVP (Utrogestan) used for luteal supplementation in cryo-warmed embryo transfer cycles. Upon consent, 224 patients women will be randomly allocated into either one of the study groups using a simple randomization method by computer-generated random numbers. Group I will receive the oral dydrogesterone, while group II will receive the vaginal microprogesterone.

ELIGIBILITY:
Inclusion Criteria:

* Normal uterine cavity
* Normal Hormonal investigation: TSH,PRL,FBS
* Frozen embryo transfer cycles: at least 2 embryos
* Primary or secondary infertility: tubal occlusion, male factor, unexplained, endometriosis, ovarian factors…
* Body mass index (BMI) ≥18 to ≤30 kg/m2

Exclusion Criteria:

* Preexisting untreated medical condition (thyroid disease, diabetes mellitus, hypertension, pulmonary conditions, cardiac condition…)
* History of three or more consecutively failed In Vitro Fertilization (IVF) cycles after embryo transfer
* History of three or more miscarriages
* Previous allergy reactions to progesterone products

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 157 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Live births per embryo transferred | until date of delivery
  Number of live births per number of embryos transferred

SECONDARY OUTCOMES:
Ongoing or Clinical pregnancy rate per started treatment cycle (CPR) | 20 weeks from Last Menstrual Period (LMP)
  The presence of a viable fetus at 20 weeks gestation or fetal heart beat on transvaginal ultrasound after 6-7 weeks of gestation
Implantation rate (IR) | 7 weeks from LMP
  Number of intrauterine gestational sacs observed on transvaginal ultrasound divided by the number of transferred embryos
Miscarriage rates | From a positive pregnancy test till 12 weeks gestation
  Pregnancy loss prior to 12 weeks of gestation
Multiple gestation rate | 6-7 weeks of gestation
  More than one intra-uterine gestation sac at 6 weeks of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon